CLINICAL TRIAL: NCT07370675
Title: Active Surveillance for Small Thyroid Nodules With Bethesda IV Cytology: A Prospective Cohort Study Protocol
Brief Title: Active Surveillance for Bethesda IV Thyroid Nodules
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Grønhøj Larsen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Christian Grønhøj Larsen, Senior registrar, PhD, DMSci, ass. prof., Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25047119
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Thyroid Cancer; Thyroid Nodule
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule | interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Surveillance (Experimental): Active surveillance with ultrasound and clinical follow-up in a 5 year period
  Interventions: Other: Active surveillance (6, 12, 18, 24, 36, 48, 60 months)

INTERVENTIONS:
Other: Active surveillance (6, 12, 18, 24, 36, 48, 60 months) — Active Surveillance og thyroid nodules with Bethesda IV cytology instead of surgery (diagnostic hemithyroidectomy).

SUMMARY:
The traditional surgical approach for Bethesda IV thyroid nodules burdens healthcare systems and patients with costs, perioperative morbidity, and potential long-term consequences of hemithyroidectomy, including hypothyroidism (requiring lifelong thyroid hormone replacement), nerve damage, infection, voice discomfort and postoperative bleeding. Moreover, patient-reported anxiety and reduced quality of life often follow surgery, regardless of benign final pathology. Conversely, surveillance strategies that include periodic ultrasound assessment, clinical examination, and patient education may reduce overtreatment, preserve thyroid function, and optimize resource utilization.

This prospective cohort protocol seeks to address these gaps by systematically evaluating the safety, feasibility, patient experience, and clinicopathologic predictors of progression for Bethesda IV nodules <2 cm managed with active surveillance.

Our hypothesis is: In patients with thyroid nodules smaller than 2 cm and cytology consistent with Bethesda IV, active surveillance is a safe and feasible alternative to immediate surgery. We hypothesize that only a minority of patients will demonstrate clinically significant tumor progression or require surgical intervention within five years, and that prospective surveillance can prevent unnecessary thyroid operations without compromising patient safety or long-term outcomes.

The primary aim of this study is to determine the proportion of patients with Bethesda IV thyroid nodules <2 cm who undergo surgical intervention or experience disease progression over a 1-, 2- and 5 year AS period.

ELIGIBILITY:
Inclusion Criteria:

* age of 30 years or older AND
* a single nodule with a Follicular neoplasm or suspicious for a follicular neoplasm (category IV in the Bethesda system) AND
* tumor size of less than 2 cm in all dimensions AND
* EU-TIRADS 3 or 4 in Ultrasound imaging examination.

Exclusion Criteria:

* EU-TIRADS 5 in Ultrasound imaging examination.
* suspicion of disseminated disease because of PET-positive lymph nodes; suspect lymph-nodes by US or by CT-scan; or signs of capsular invasion of the tumor, or irregular shape or margins, extrathyroidal growth OR
* tumor placement at a high-risk location (in the thyroid capsule with extracapsular extension toward vessels, RLN, or the trachea) OR
* previous thyroid surgery OR
* concomitant hyperparathyroidism (ionized calcium > 1.32 mmol/L and PTH > 6 pmol/L) OR
* if the patient is pregnant OR
* If the patient is unable to give informed consent. OR
* If calcitonin is elevated above normal level

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2033-01-16 (Estimated); Study Completion 2033-01-16 (Estimated)

PRIMARY OUTCOMES:
Number of participants who undergo surgical intervention or experience disease progression during active surveillance | From enrollment in to active surveillance to the end of the follow-up programe at 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Otolaryngology, Head and Neck SurgeryRigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No